CLINICAL TRIAL: NCT05069116
Title: The Impact of Covid 19 Pandemic on the Training of General Surgery Residents
Status: Completed | Type: Observational
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Calin Popa, Principal Investigator, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: SURG TRAINING - COVID
Record Dates: First submitted 2021-10-05; First posted 2021-10-06 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: COVID-19 Pandemic; Educational Problems
MeSH Terms: conditions — COVID-19 | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pre-Covid era
  Interventions: Other: Training in surgery
- Covid-era
  Interventions: Other: Training in surgery

INTERVENTIONS:
Other: Training in surgery — The study evaluates the training process of general surgery residents - in classic surgery, as well as laparoscopic surgery, from hospital activity to extracurricular activities.

SUMMARY:
The educational process of general surgery residents is a very important step in every surgeon's career, which is often overlooked or neglected. The Covid-19 pandemic has inflicted deep changes in the medical activity in general and in the training process of young doctors in particular.

Our study aims to assess the impact of the Covid-19 pandemic on the educational process of general surgery residents, through a comparative study. The responses of resident doctors at a questionnaire, in two different time periods, will be compared: pre-Covid era (December 2019) and Covid era (December 2020).

ELIGIBILITY:
Inclusion Criteria:

* General surgery residents
* Above second year of residency
* Residency program in Cluj-Napoca Medical Centre

Exclusion Criteria:

* Incomplete responses to the questionnaire
* Refusal to be included in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: general surgery resident doctors
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
The impact of the pandemic on the educational process | December 2019-December 2020
  Active participation in the operating room (hours/day, day/week), Theoretical education (hours/week), possibilities of extracurricular training

CONTACTS AND LOCATIONS:
Locations (1):
- "Iuliu Haţieganu" University of Medicine and Pharmacy, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Undecided